CLINICAL TRIAL: NCT00767351
Title: Intraindividual Variation of Serum Metformin in a Cohort of Patients With Type 2 DM and Moderately Reduced Renal Function
Brief Title: Variation in Serum Levels of Metformin in Patients With Reduced Renal Function
Status: Completed | Type: Observational
Sponsor: Skane University Hospital (Other)
Responsible Party: Principal Investigator, Gunnar Sterner, PhD, Skane University Hospital
Other Study IDs: 001
Record Dates: First submitted 2008-10-06; First posted 2008-10-07 (Estimated); Last update posted 2018-09-10 (Actual); Status verified 2018-09

CONDITIONS: Diabetes Mellitus Type 2; Metformin; Pharmacokinetics
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Metformin is widely used for treatment of type 2 diabetes mellitus. Side-effects are few and mainly from the gastrointestinal tract. Since metformin is cleared from the blood exclusively via the kidneys reduced renal function is a relative contraindication. We have earlier demonstrated that metformin safely can be used to a lower GFR level of 30 ml/min/1.73. Below that level the risk of lactacidosis, a severe complication, increases.

In the present study we plan to analyse serum levels of metformin repeatedly in patients with moderate renal failure (CKD = GFR of 30-60 ml/min/1.73). Blood samples will be taken as trough values in the morning, week 0, 2, 4, and 8 and at four weeks a blood sample will be taken two hours after intake of the morning dose of metformin. Renal function will be estimated with creatinine and cystatin C at each occasion. The intraindividual variation of metformin will be calculated.

The study rests on a new method for measuring metformin. The technique uses Liquid Chromatography Tandem Mass Spectometry (LCMSMS). Proteins are removed from serum by adding acetonitrile to the sample. After centrifugation a diluted portion of the supernatant is injected into the LCMSMS-system. The total runtime for a sample is 6 minutes.

The study will show if variation in serum levels of metformin measured in the same patient is high or low and thus give us better understanding whether a change i serum level is due to biological variation or to increased retention caused by progressive renal failure.

ELIGIBILITY:
Inclusion Criteria:

* Patients above the age of 18 years with type 2 diabetes mellitus.
* Reduced renal function measured as estimated GFR (below 60 ml/min/1.73).
* Treatment with metformin on going.

Exclusion Criteria:

* Severely reduced GFR (< 30 ml(min/1.73)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with type 2 DM followed at the out-patient department at the hospital will be asked to join the study
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2008-10; Primary Completion 2009-06 (Actual); Study Completion 2009-07 (Actual)

REFERENCES:
- [Derived] Frid A, Sterner GN, Londahl M, Wiklander C, Cato A, Vinge E, Andersson A. Novel assay of metformin levels in patients with type 2 diabetes and varying levels of renal function: clinical recommendations. Diabetes Care. 2010 Jun;33(6):1291-3. doi: 10.2337/dc09-1284. Epub 2010 Mar 9. PMID 20215446